CLINICAL TRIAL: NCT01822470
Title: Small Intestinal Bacterial Overgrowth: A Prospective Registry
Acronym: SIBO
Status: Enrolling by invitation | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Progenity, Inc. (Industry)
Responsible Party: Principal Investigator, John M. Wo, Professor of Medicine, Indiana University
Other Study IDs: 1209009531
Record Dates: First submitted 2013-03-25; First posted 2013-04-02 (Estimated); Last update posted 2025-03-03 (Actual); Status verified 2024-08

CONDITIONS: Functional Dyspepsia; Small Intestinal Bacterial Overgrowth
Keywords: functional dyspepsia; post prandial distress syndrome; small bowel bacteria overgrowth; epigastric pain syndrome; diarrhea; bloating; post prandial fullness; weight loss
MeSH Terms: conditions — Diarrhea; Weight Loss

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — DNA will be kept from patients jejunal aspirate and mucosal biopsy. In addition, patient serum will be kept
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Study group: a. Study Subjects will be recruited from patients who are already undergoing upper enteroscopy and aspiration for diagnosis of SIBO.
- Control group: b. Control Subjects will be recruited from patients who are already undergoing a double balloon enteroscopy or upper enteroscopy for another medical reason

SUMMARY:
The purpose of this study is to investigate the prevalence of small intestinal bacterial overgrowth (SIBO) in patients who will be undergoing an enteroscopy as an outpatient procedure with symptoms of functional dyspepsia. In addition, the investigators would like to identify the types of bacteria that are present in the small intestines in patients with SIBO and compare two different diagnostic tools: microbiologic culture and DNA sequencing of bacteria.

The aim is to compare the microbiota between patients with and without the clinical complications of SIBO

DETAILED DESCRIPTION:
Same as above

ELIGIBILITY:
1.Study Subjects Inclusion Criteria i. All patients who are undergoing small bowel aspiration for suspected SIBO regardless etiology.

Exclusion Criteria i. Use of colon cleansing prep in the past 1 month ii. Treatment with antibiotics in the past 30 days (antibiotics are allowable for patients undergoing clinical indicated repeat aspiration to determine bacteria clearance) iii. Use of probiotics in the past 30 days iv. Contraindication for upper endoscopy for any reason v. Prisoners vi. Pregnant vii. Unable to give own informed consent

2 Control Subjects Inclusion Criteria i. Patients who are undergoing double balloon enteroscopy or upper enteroscopy for another medical reason.

Exclusion Criteria i. Diagnosis of SIBO ii. Diagnosis of functional dyspepsia iii. Established risk factors for SIBO (ANY of the following)

1. Connective tissue disorder (scleroderma, polymyositis, mixed connective tissue disease, or systemic lupus
2. Resection of ileocecal valve for any reason
3. Chronic intestinal pseudo-obstruction
4. Small bowel blind limb, diverticulum or fistula
5. Surgery with decreased gastric acid exposure for small bowel a. Gastric surgery with vagotomy (Bilroth I, Bilroth II, vagotomy/pyloroplasty) or gastric bypass iv. Use of colon cleansing prep in the past 1 month v. Use of antibiotics in the past 30 days vi. Use of probiotics in the past 30 days vii. Contraindication for upper endoscopy for any reason viii. Prisoners ix. Pregnant x. Unable to give own informed

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: a. All adult patients who are undergoing small bowel aspiration for suspected SIBO regardless etiology
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-01-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To determine the predictors for SIBO in patients with functional dyspepsia, who do not have the established risk factors for SIBO | two years
  In this population, prevalence of potential predictors of SIBO will be compared between subjects with and without a diagnosis of Gram Negative Bacteria SIBO

SECONDARY OUTCOMES:
A registry of patients undergoing proximal jejunal aspiration for suspected small intestinal bacterial overgrowth | Two years
  A prospective registry will be created for all subjects who are undergoing jejunal aspirate for clinical indications. Private health information will be excluded from the data registry. Data collected for the registry will include:
  1. Demographics
  2. Patient Assessment of Gastrointestinal Disorders-Symptom Severity Index total and subscale scores
  3. Presence of functional gastrointestinal disorders
  4. Established risk factors of gram negative small intestinal bacterial overgrowth.
  5. Established risk factors of upper respiratory tract small intestinal bacterial overgrowth
The demographics, clinical history, and symptoms in patients with and without SIBO | One day
  Demographics 2. Patient Assessment of Gastrointestinal Disorders-Symptom Severity Index total and subscale scores 3. Presence of functional gastrointestinal disorders 4. Established risk factors of gram negative small intestinal bacterial overgrowth.
  5. Established risk factors of upper respiratory tract small intestinal bacterial overgrowth
Characterize the clinical differences between small intestinal bacterial overgrowth by upper respiratory tract bacteria and small intestinal bacterial overgrowth by gram-negative bacilli bacteria | One day
  clinical differences between small intestinal bacterial overgrowth by upper respiratory tract bacteria
Compare the composition between luminal and mucosal bacteria in the proximal small bowel | One day
  Compare the results of bacteria species isolated from molecular polymerase chain reaction identification between luminal aspiration samples and mucosa biopsy samples.

CONTACTS AND LOCATIONS:
Overall Officials: John Wo, MD, Principal Investigator — Indiana University Hospital
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided